CLINICAL TRIAL: NCT03115424
Title: Effect of GLP-1 Receptor Agonism on Weight and Caloric Intake in Subjects After Sleeve Gastrectomy
Brief Title: Effect of GLP-1 Receptor Agonism After Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16-004253
Record Dates: First submitted 2017-04-05; First posted 2017-04-14 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Obesity
Keywords: Weight Loss; Bariatric Surgery
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sleeve Gastrectomy Placebo (Placebo Comparator): Subjects undergoing Sleeve Gastrectomy (SG) will be randomized 1:1 at the time of 3 month visit after bariatric surgery.
  Interventions: Drug: Placebos
- Sleeve Gastrectomy Saxenda (Active Comparator): Subjects undergoing Sleeve Gastrectomy (SG) will be randomized 1:1 at the time of 3 month visit after bariatric surgery.
  Interventions: Drug: Saxenda
- RYGB (Sham Comparator): Twenty five subjects will be recruited from the Nutrition Clinic at Mayo Clinic Rochester prior to undergoing RYGB surgery.
  Interventions: Procedure: RYGB

INTERVENTIONS:
Drug: Saxenda — Saxenda is a glucagon-like peptide-1 (GLP-1) receptor agonist indicated as an adjunct to a reduced calorie diet and increased physical activity for chronic weight management in adult patients. Subjects will be recruited and screened prior to undergoing bariatric surgery. Subjects undergoing SG will be randomized 1:1 at month 3 post surgery to Saxenda, 0.6mg SQ daily, with weekly titration of 0.6mg until maintenance dose of 3mg/daily reached. Subjects will remain on study drug for duration of study (33 months). After undergoing surgery, study visits will be timed to coincide with the standard clinical follow-up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.
  Other Names: Liraglutide
  Arms: Sleeve Gastrectomy Saxenda
Drug: Placebos — Subjects will be recruited and screened prior to undergoing bariatric surgery.Subjects undergoing SG will be randomized 1:1 at months 3 post surgery to Placebo, 0.6mg SQ daily, with weekly titration of 0.6mg until maintenance dose of 3mg/daily reached. Subjects will remain on study drug for duration of study (33 months). After undergoing surgery, study visits will be timed to coincide with the standard clinical follow-up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.
  Other Names: Placebo for Saxenda (Liraglutide)
  Arms: Sleeve Gastrectomy Placebo
Procedure: RYGB — Subjects will be recruited and screened prior to undergoing bariatric surgery. After undergoing surgery, study visits will be timed to coincide with the standard clinical follow-up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.
  Arms: RYGB

SUMMARY:
Observational studies suggest that bariatric surgery is the most effective intervention for weight loss. Comparative effectiveness of Roux-en-Y Gastric Bypass (RYGB) and Sleeve Gastrectomy (SG) demonstrate that RYGB is significantly superior to SG in terms of weight loss and glycemic control. Both RYGB and SG increase GLP-1 concentrations which directly affect B-cell function. Data has shown that the postprandial rise in GLP-1 might affect feeding behavior after RYGB and to a lesser extent SG, where the increase in GLP-1 is less marked. In this study the investigators propose to randomize subjects undergoing SG to receive either placebo or Liraglutide, a GLP-1 receptor agonist, to compare weight loss and CV risk factors.

DETAILED DESCRIPTION:
A total of 75, non diabetic adults, scheduled for bariatric surgery at Mayo Clinic Rochester, will be enrolled. Of these, 25 will be scheduled for Roux-en-Y Gastric Bypass surgery (RYGB), while the remainder (50) will be scheduled for Sleeve Gastrectomy (SG). The study team will play no role in assignment of the surgical procedure. Following surgery, at month 3, subjects undergoing SG will be randomized to either Saxenda or placebo, subcutaneously once daily. Subjects randomized to Saxenda or placebo will take for the duration of the study (33 months). Follow up study visits for all subjects will be timed to coincide with the standard clinical follow up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-65 years of age
2. Seen at Mayo Clinic Nutrition Clinic and have received authorization for bariatric surgery.
3. No active physical illness which will interfere with mobility or weight loss after bariatric surgery.
4. Females who are sexually active and able to become pregnant must agree to use birth control for duration of study if randomized to Saxenda/Placebo.

Exclusion Criteria:

1. Prior use of glucose lowering medication in the 3 months prior to screening.
2. A fasting glucose ≥ 126mg/dl or an HbA1c ≥ 6.5% will be taken as evidence of type 2 diabetes and therefore patients will be deemed ineligible for participation.
3. Prior abdominal surgery other than cholecystectomy, appendectomy or hysterectomy.
4. Pregnancy or active consideration of pregnancy during the period of study. Subjects will be discontinued if they become pregnant during the study.
5. Hypersensitivity to liraglutide or any product components.
6. Personal or family history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia type 2.
7. Prior history of pancreatitis, cholelithiasis or cholecystitis.
8. Concurrent use of insulin or any other GLP-1 receptor agonist.
9. Active, severe psychiatric disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleeve Gastrectomy Saxenda: Subjects underwent Sleeve Gastrectomy (SG) were randomized 1:1 at the time of 3 month visit after bariatric surgery.
  Saxenda: Saxenda is a glucagon-like peptide-1 (GLP-1) receptor agonist indicated as an adjunct to a reduced calorie diet and increased physical activity for chronic weight management in adult patients. Subjects were recruited and screened prior to undergoing bariatric surgery. Subjects undergoing SG will were randomized 1:1 at month 3 post surgery to Saxenda, 0.6mg SQ daily, with weekly titration of 0.6mg until maintenance dose of 3mg/daily reached. Subjects will remain on study drug for duration of study. After undergoing surgery, study visits were timed to coincide with the standard clinical follow-up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.
- Sleeve Gastrectomy Placebo: Subjects underwent Sleeve Gastrectomy (SG) were randomized 1:1 at the time of 3 month visit after bariatric surgery.
  Placebos: Subjects were recruited and screened prior to undergoing bariatric surgery. Subjects undergoing SG were randomized 1:1 at months 3 post-surgery to Placebo, 0.6mg SQ daily, with weekly titration of 0.6mg until maintenance dose of 3mg/daily reached. Subjects remained on study drug for duration of study. After undergoing surgery, study visits were timed to coincide with the standard clinical follow-up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.
- Roux-en-Y Gastric (RYGB): Subjects were recruited from the Nutrition Clinic at Mayo Clinic Rochester prior to undergoing RYGB surgery.
  RYGB: Subjects were recruited and screened prior to undergoing bariatric surgery. After undergoing surgery, study visits were timed to coincide with the standard clinical follow-up visits at months 3, 6, 9, 12, 18, 24, 30 and 36.
Period: Overall Study
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB)
Started | 12 | 9 | 25
Completed | 12 | 9 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB) | Total
Number analyzed (Participants) | 12 | 9 | 25 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12) | 46 (11) | 42 (9) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 22 | 40
  Male | 2 | 1 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Subjects calculated weight in kilograms
Time Frame: baseline and 36 months
Population: Data was not collected nor analyzed for eight subjects in the Sleeve Gastrectomy Saxenda arm. Data was not collected nor analyzed for seven subjects in the Sleeve Gastrectomy Placebo arm. Data was not collected nor analyzed for thirteen subjects in the Roux-en-Y Gastric (RYGB).
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB)
Number analyzed (Participants) | 12 | 9 | 25
kilograms
  baseline | 127 (7) | 130 (8) | 126 (4)
  36 months: number analyzed (Participants) | 4 | 2 | 12
  36 months | 75 (8) | 107 (10) | 98 (7)

2. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (top number of blood pressure reading)
Time Frame: baseline and 36 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Millimeters of Mercury
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB)
Number analyzed (Participants) | 12 | 9 | 25
Millimeters of Mercury
  baseline | 129 (4) | 130 (7) | 123 (4)
  36 months: number analyzed (Participants) | 4 | 2 | 12
  36 months | 112 (7) | 128 (1) | 122 (7)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure (bottom number of blood pressure reading)
Time Frame: baseline and 36 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Millimeters of Mercury
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB)
Number analyzed (Participants) | 12 | 9 | 25
Millimeters of Mercury
  baseline | 86 (3) | 83 (6) | 76 (2)
  36 months: number analyzed (Participants) | 4 | 2 | 12
  36 months | 84 (4) | 93 (13) | 82 (3)

4. Secondary Outcome: Low-density Lipoprotein (LDL)
Description: LDL's carry cholesterol through the bloodstream. LDL is called bad cholesterol because high amounts can form plaques in the blood vessels, increasing risk for heart disease. Adult normal range is less than 100 mg/dL.
Time Frame: baseline and 36 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB)
Number analyzed (Participants) | 12 | 9 | 25
mg/dL
  baseline | 114 (9) | 101 (11) | 99 (5)
  36 months: number analyzed (Participants) | 4 | 2 | 12
  36 months | 106 (20) | 68 (1) | 90 (7)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 36 months
Arm/Group | Sleeve Gastrectomy Saxenda | Sleeve Gastrectomy Placebo | Roux-en-Y Gastric (RYGB)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/9 | 0/25
Other Adverse Events (participants affected / at risk) | 2/12 | 1/9 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleeve Gastrectomy Saxenda (N=12) | Sleeve Gastrectomy Placebo (N=9) | Roux-en-Y Gastric (RYGB) (N=25)
Seizure (Nervous system disorders) | 1 (2) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleeve Gastrectomy Saxenda (N=12) | Sleeve Gastrectomy Placebo (N=9) | Roux-en-Y Gastric (RYGB) (N=25)
Hgb < 11.5 g/dL (Blood and lymphatic system disorders) | 0 | 0 | 1 (1)
Nausea (General disorders) | 2 (2) | 1 (1) | 14 (14)
Vomiting (General disorders) | 2 (2) | 1 (1) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03115424/Prot_SAP_001.pdf